CLINICAL TRIAL: NCT04650451
Title: A Phase 1/2, Open-Label, Multicenter, Non-Randomized, Safety and Activity Study of HER2-Targeted Dual Switch CAR-T Cells (BPX-603) In Subjects With Previously Treated Advanced HER2-Positive Solid Tumors
Brief Title: Safety and Activity Study of HER2-Targeted Dual Switch CAR-T Cells (BPX-603) in Subjects With HER2-Positive Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a Dose Limiting Toxicity in another sister trial with same technology.
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPX603-201A
Record Dates: First submitted 2020-11-20; First posted 2020-12-02 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: HER-2 Gene Amplification; HER2-positive Gastric Cancer; HER2-positive Breast Cancer; HER-2 Protein Overexpression; Solid Tumor, Adult
Keywords: HER2; CAR-T; breast cancer; solid tumors; gastric cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Receptors, Chimeric Antigen; Automobiles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HER2-targeted dual-switch CAR-T cells (Experimental): Subjects will receive one dose of BPX-603 on Day 1, followed by rimiducid IV infusion weekly (as tolerated) starting on Day 8 and continued until treatment discontinuation criteria are met.
  Interventions: Biological: chimeric antigen receptor (CAR) T cell therapy

INTERVENTIONS:
Biological: chimeric antigen receptor (CAR) T cell therapy — HER2-targeted dual-switch CAR-T cells
  Other Names: CAR-T; BPX-603; autologous CAR-T

SUMMARY:
This is a Phase 1/2, open-label, multicenter, non-randomized study to investigate the safety, tolerability, and clinical activity of HER2-specific dual-switch CAR-T cells, BPX-603, administered with rimiducid to subjects with previously treated, locally advanced or metastatic solid tumors which are HER2 amplified/overexpressed.

DETAILED DESCRIPTION:
* Phase 1: Cell dose escalation to identify the maximum dose of BPX-603 administered without or with rimiducid. The first subject in each dose cohort will receive BPX-603 alone (without rimiducid) in order to assess safety of the CAR-T monotherapy.
* Phase 2: Indication-specific dose expansion to assess the safety, pharmacodynamics (including BPX-603 persistence and response to temsirolimus as applicable), and clinical activity at the recommended dose for expansion (RDE) identified in Phase 1 in various HER2+ solid tumors.
* During Phase 1 or 2, temsirolimus (single IV dose at 25 mg) may be administered following BPX-603 infusion in response to treatment-emergent toxicity in order to activate the iRC9 safety switch.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of HER2 amplification/overexpression by local testing.
* Histologically or cytologically confirmed diagnosis of a locally advanced unresectable or metastatic HER2+ solid tumor malignancy for which standard treatment is no longer effective, does not exist, or subject is ineligible.
* Subjects with a solid tumor malignancy for which HER2-targeted therapy is approved as a standard treatment (e.g., breast, gastric cancers) must have received prior treatment with approved HER2-directed therapy.
* Measurable disease (at least one target lesion) per RECIST v1.1.
* Life expectancy > 12 weeks.
* ECOG 0-1.
* Adequate organ function.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system metastases.
* Prior CAR T cell or other genetically-modified T cell therapy.
* Impaired cardiac function or clinically significant cardiac disease.
* Symptomatic intrinsic lung disease or those with extensive tumor involvement of the lungs.
* Severe intercurrent infection.
* Pregnant or breastfeeding.
* Known HIV positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects experiencing Dose Limiting Toxicities at increasing doses of BPX-603 | 35 days from time of BPX-603 infusion
  Dose limiting toxicities are defined as BPX-603-related adverse events.
Maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) | through Phase 1 completion, up to 2 years
  Identify the optimal dose of BPX-603 for Phase 2.

SECONDARY OUTCOMES:
Persistence of HER2-CAR T cells (cell counts) | measured over time from baseline through study completion, up to 5 years
  The persistence over time of BPX-603 CAR T cells in the peripheral blood as determined by flow cytometry (% CAR+ cells).
Expansion of HER2-CAR T cells (vector copy number) | measured over time from baseline through study completion, up to 5 years
  The expansion over time of BPX-603 CAR T cells in the peripheral blood as determined by qPCR (copies/ug gDNA).
Antitumor activity of BPX-603 | through study completion, up to 5 years
  Overall response rate

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego (UCSD), La Jolla, California
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas